CLINICAL TRIAL: NCT04623203
Title: The Prognosis of Migraine and Tension-Type Headache in Children and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Jacob.genizi, Manager pediatric neurology unit, Bnai Zion Medical Center
Other Study IDs: BNZ 109-18
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Children, Only; Headache, Migraine; Headache, Tension
Keywords: Headache; Migraine; Tension Type Headache; Adolescents; Outcome
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children with migraine: Children that were diagnosed at the neurology clinic with migraine at the years 2007-2010. A follow up visit at 2020 of their current headache condition.
  Interventions: Other: No intervention
- children with TTH: children that were diagnosed at the neurology clinic with TTH at the years 2007-2010. A follow up visit at 2020 of their current headache condition.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Children and adolescents that visited the pediatric neurology clinic at the Bnai Zion medical center do to migraine or TTH headache between the years 2007-2010 were reevaluated. We used a structured headache questionnaire through a phone interview with the patients and their caregivers. Data regarding demographics, the patients' and families' medical history, and headache history, past and current (age at onset, location, quality, frequency, duration of episodes, aura, associated symptoms and treatment) were collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine or TTH headache according to the ICHD-3 criteria.
* Can describe the current headache status.

Exclusion Criteria:

* Secondary headaches.

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents that visited the pediatric neurology clinic at the Bnai Zion medical center do to migraine or TTH headache between the years 2007-2010
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Headache diagnosis according to the ICHD-3 criteria | 10 years from initial diagnosis
  The diagnosis of headache episodes at follow-up according to the ICHD-3 criteria; either Migraine or TTH.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob GENIZI, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Not yer decided how